CLINICAL TRIAL: NCT07286409
Title: Nebulized Furosemide, Heparin, Hypertonic Saline in Mechanically Ventilated Acute Respiratory Distress Syndrome Adult Patients: A Randomized Controlled Clinical Trial
Brief Title: Nebulized Furosemide, Heparin, Hypertonic Saline in Mechanically Ventilated Acute Respiratory Distress Syndrome Adult Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: nebulized drugs in ARDS
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Distress Syndrome; Mechanical Ventilation Complication
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- frusemide (Active Comparator): The furosemide group will receive 40 mg furosemide in 4 ml of 0.9% saline, administered /6 hours for 7 days
  Interventions: Drug: nebulization
- heparin (Active Comparator): The heparin group will receive inhaled unfractionated heparin at a dose of 10,000 in 4 ml of 0.9% saline IU/6 h daily for 7 days via ventilator circuit.
  Interventions: Drug: nebulization
- hypertonic saline (Active Comparator): This group will receive inhaled hypertonic saline 3% in a dose of 4ml /6 h daily for 7 days.
  Interventions: Drug: nebulization
- control (Placebo Comparator): This group will receive inhaled normal saline 0.9 % in a dose of 4ml /6 h daily for 7 days.
  Interventions: Drug: nebulization

INTERVENTIONS:
Drug: nebulization — Study solutions will be administered via a vibrating mesh nebulizer (Aerogen® Pro, Aerogen Ltd, Ireland) placed at the Y-piece of the ventilator circuit, proximal to the patient. The nebulizer will be used with its specific T-piece adapter. The nebulizer will be placed at the Y-piece (proximal to the patient), between the endotracheal tube and the circuit. To optimize aerosol delivery, a standardized nebulization protocol will be followed. For the 30-minute duration of each treatment, the ventilator will be set to Volume Control or Assist-Control mode with a constant inspiratory flow of 40-50 L/min, an inspiratory-to-expiratory ratio of 1:3, and an end-inspiratory pause of 0.5 seconds. The heated humidifier will be turned off 15 minutes before and bypassed during the nebulization period. Immediately after the 30-minute nebulization is complete, the humidification chamber will be reconnected, and the heated humidifier will be turned back on.

SUMMARY:
There are no specific drugs or therapies available to directly treat/prevent ARDS. Mechanical ventilation with an aim to minimize Ventilator Induced Lung Injury (VILI) and management of refractory hypoxemia are the keystones in supportive management of ARDS.

DETAILED DESCRIPTION:
Furosemide: Nebulized furosemide has been studied as a potential treatment option for ARDS patients due to its diuretic properties and potential to reduce pulmonary edema. Research on the effectiveness of furosemide nebulization in ARDS patients could provide valuable insights into its potential role in managing respiratory distress and improving outcomes. Furosemide may reduce pulmonary edema via diuretic and anti-inflammatory effects.

Heparin: Nebulized heparin has been proposed as a treatment for ARDS patients due to its anti-inflammatory and anticoagulant effects. By investigating the effectiveness of heparin nebulization in reducing pulmonary inflammation and improving oxygenation in ARDS patients, clinicians can gain a better understanding of its therapeutic potential in this critical condition. - ARDS involves fibrin deposition in alveoli, worsening compliance. Heparin may reduce microthrombosis and inflammation (anti-TNF-α effects).

Hypertonic saline: Nebulized hypertonic saline has been suggested as a potential therapy for ARDS patients due to its ability to reduce airway inflammation and improve mucociliary clearance. Examining the effectiveness of hypertonic saline nebulization in ARDS patients could offer valuable insights into its impact on respiratory function and recovery in this challenging patient population. Hypertonic saline may improve mucus clearance and alveolar fluid absorption.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* ICU admission, mechanical ventilation for < 7 days
* ARDS diagnosed within 24 hours per the Berlin Definition, which includes Chest x-ray showing bilateral opacities, not fully explained by effusions, lung collapse; Respiratory failure not fully explained by cardiac failure or fluid overload, and exclusion of hydrostatic edema (by echocardiography);
* Oxygenation and ventilator settings matching one of the three categories of ARDS: Mild: 200 mmHg < PaO2/FIO2 ≤ 300 mmHg with positive end-expiratory pressure (PEEP) or continuous positive airway pressure (CPAP) ≥ 5 cm H2O. Moderate: 100 mm Hg < PaO2/FIO2 ≤ 200 mm Hg with PEEP ≥ 5 cm H2O. Severe: PaO2/FIO2 ≤ 100 mm Hg with PEEP ≥ 5 cm H2O.

Exclusion Criteria:

* 1- Pregnant Patient. 2- Refusal to participate in the trial by the patient's guardian. 3- Known allergy to furosemide or heparin. 4- Active major bleeding, recent intracranial hemorrhage 5- End-stage renal disease 6- Severe chronic liver disease. 7- Uncontrolled shock (e.g., high vasopressor doses). 8- Advanced directives limiting care (e.g., do-not-resuscitate orders), which could affect mortality outcomes.

  9- Body Mass Index (BMI) > 40 or severe obesity, which can severely impact lung mechanics and confound results.

  10- Electrolyte imbalance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Murray Lung Injury Score | in the morning of 7 days of mechanical ventillation
  Murray lung injury score will be calculated daily in the morning (8:00 am) based on information obtained from:
  1. Number of quadrants of infiltrations from chest X-ray.
  2. Hypoxic index.
  3. Positive end expiratory pressure (PEEP (cmH2O)) required on the ventilator to get better oxygenation.
  4. Static compliance will be calculated daily in the morning (8:00 am) based on information obtained from:
  a) Number of quadrants of infiltrations from chest X-ray. b) Hypoxic index. c) Positive end expiratory pressure (PEEP (cmH2O)) required on the ventilator to get better oxygenation.
  d) Static compliance

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Tanta university, Tanta, El Gharbyia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided